CLINICAL TRIAL: NCT05316441
Title: The Effect of Achievement Skill Development Psychoeducation Based on Positive Psychotherapy in Adolescents on Achievement Motivation
Brief Title: Positive Psychotherapy in Adolescents on Achievement Motivation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Eda Albayrak, Research Assistant, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Erciyes Universty
Record Dates: First submitted 2022-03-15; First posted 2022-04-07 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Adolescent Behavior
MeSH Terms: conditions — Adolescent Behavior

STUDY DESIGN:
Intervention Model Description: The research was designed in an experimental model with an intervention-control group. The sample of the research; It consists of 60 students (30 controls, 30 experiments) with 80% power, 95% confidence interval and 0.05 margin of error.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): A total of 5 sessions of 1.5 hours of group therapy will be applied to the Intervention Group. Group therapies will be carried out over the internet once a week, after appropriate days and times are determined.
  Interventions: Behavioral: psychoeducation
- Control Group (No Intervention): The control group will not be interfered with.

INTERVENTIONS:
Behavioral: psychoeducation — Positive Psychotherapy is a recently emerged therapy method that works on talents. In the study, success skill development psychoeducation based on positive psychotherapy will be applied.
  Arms: Intervention Group

SUMMARY:
The aim of this study is to determine the effect of success skill development psychoeducation based on Positive Psychotherapy on the achievement motivation of adolescents.

DETAILED DESCRIPTION:
The foundation of positive psychotherapy (PPT) Prof. Dr. It was cast by Nossrat Peseschkian. Psychodynamic approaches, existential-humanistic approaches, cultural therapy approaches and behavioral approaches are used in therapy. Positive Psychotherapy states that people have two basic abilities, namely loving and knowing.

In line with the ability to love, primary abilities (love, modeling, relationship/contact, time, patience, trust, belief/religion, doubt, certainty, sexuality, hope and integrity) are formed; In line with the ability to know, secondary abilities (punctuality, orderliness, cleanliness, obedience, courtesy, honesty, loyalty, justice, hard work/success, frugality and reliability) are formed, which are behavioral categories.

These real abilities develop with family, society, environment and time and become the character of the person, and the degree of whether or not the real abilities are in the person plays a decisive role in both the individual's own mental state and interpersonal relations. The ability to succeed, which is one of the secondary abilities, is extremely important for people to have goals and passions in life.

The two most important components of a successful learning-teaching process are providing learner motivation and ensuring the learner's behavioral, sensory and cognitive participation in this process.

Considering that a significant decrease in achievement motivation is observed especially in adolescents with advancing age, the achievement motivation levels of learners against course processes emerge as an important requirement.

ELIGIBILITY:
Inclusion Criteria:

Being a high school student. Having equipment and internet to attend group sessions. Volunteer to work.

Exclusion Criteria:

Not having the equipment and internet to attend group sessions. Not being willing to work.

Ages: 15 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2022-04 (Estimated); Primary Completion 2022-05 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Achievement Motivation | Change = Pre-psychoeducational assessment (Time 1), immediately after psychoeducation (Time 2).
  The scale consists of 9 items and two sub-dimensions. Of these dimensions, there are 2 items in the expectation sub-dimension and 6 items in the value sub-dimension. The lowest score that can be obtained from the scale is 8, and the highest score is 40.

IPD SHARING:
Plan to Share IPD: Undecided